CLINICAL TRIAL: NCT01311336
Title: Randomized Phase II Pilot Study of Loratadine for the Prevention of Pain Caused by the Granulocyte Colony Stimulating Factor Pegfilgrastim
Brief Title: Evaluation of Loratadine for Prevention of Pegfilgrastim-Induced Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Collaborators: Cancer and Leukemia Group B (Network)
Responsible Party: Principal Investigator, Steven Grunberg, Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: VCC 1012
Record Dates: First submitted 2011-03-08; First posted 2011-03-09 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Pegfilgrastim-induced Back and Leg Pain
Keywords: Pegfilgrastim; Loratadine; Myalgia/arthralgia
MeSH Terms: conditions — Myalgia; Arthralgia | interventions — Loratadine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Loratadine (Active Comparator): Loratadine 10 mg once a day for 7 days beginning the day of pegfilgrastim treatment in patients with pegfilgrastim-induced back and leg pain during the previous treatment cycle
  Interventions: Drug: Loratadine
- Placebo (Placebo Comparator): Placebo once a day for 7 days beginning the day of pegfilgrastim treatment in patients with pegfilgrastim-induced back and leg pain during the previous treatment cycle
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Loratadine — loratadine 10 mg capsule orally once daily for 7 days beginning the day of administration of pegfilgrastim
  Other Names: Claritin
  Arms: Loratadine
Drug: placebo — placebo capsule orally once daily for 7 days beginning the day of administration of pegfilgrastim
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the incidence of pegfilgrastim-induced back and leg pain and to determine whether the antihistamine loratadine can prevent pegfilgrastim-induced back and leg pain.

DETAILED DESCRIPTION:
Pegfilgrastim is a myeloid growth factor that stimulates neutrophil precursors and can be used to decrease infection risk associated with neutropenia. However pegfilgrastim may induce back and leg pain in 20-50% of patients. No intervention has been consistently successful in treating or preventing this pain.

The exact mechanism of pegfilgrastim-induced pain is unknown but may be related to histamine-mediated inflammation. Several case reports and anecdotal reports have suggested efficacy of antihistamines for this indication.

This study will have two parts. In the first part (Observational Phase), patients receiving pegfilgrastim will be surveyed to document the incidence of significant pegfilgrastim-induced back and leg pain. In the second part (Treatment Phase), patients who previously experienced such pain will be randomized to receive a 7-day course of either the antihistamine loratadine or placebo to determine whether pegfilgrastim-induced back and leg pain can be prevented with this intervention.

ELIGIBILITY:
Inclusion Criteria:

* histologic or cytologic evidence of malignancy
* scheduled to receive pegfilgrastim with two consecutive cycles of similar chemotherapy with at least a 14 day interval between cycles
* adequate renal function: estimated creatinine clearance > 30 ml/min
* adequate hepatic function: AST, ALT, total bilirubin <= 2.5 x ULN
* age >= 18 years
* performance status 0-3
* able to read and understand English
* signed Informed Consent

Exclusion Criteria:

* history of hypersensitivity or intolerance to antihistamines
* concurrent use of antihistamines other than study medications during or for 2 days prior to the study period except for a single dose of antihistamine as required for administration of chemotherapy or blood transfusion
* concomitant use of amiodarone
* previous use of pegfilgrastim or filgrastim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2011-05; Primary Completion 2013-06 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Prevention of pegfilgrastim-induced back and leg pain by administration of the antihistamine loratadine | one week after pegfilgrastim
  Patients who experience significant pegfilgrastim-induced back and leg pain during the first cycle of pegfilgrastim therapy are randomized to receive loratadine or placebo during the second cycle of pegfilgrastim therapy

SECONDARY OUTCOMES:
Identification of adverse events when loratadine is given to prevent pegfilgrastim-induced back and leg pain | one week after pegfilgrastim
  Adverse events will be recorded for patients receiving loratadine or placebo to prevent pegfilgrastim-induced back and leg pain
Incidence of pegfilgrastim-induced back and leg pain | One week after pegfilgrastim
  Patients receiving pegfilgrastim for the first time will be surveyed to document the incidence of significant pegfilgrastim-induced back and leg pain

CONTACTS AND LOCATIONS:
Overall Officials: Steven M Grunberg, MD, Study Chair — University of Vermont
Locations (7):
- United States (7):
  - Cancer Care of Maine, Brewer, Maine
  - Maine Center for Cancer Medicine, Scarborough, Maine
  - York Hospital, York Village, Maine
  - CR Wood Cancer Center, Glens Falls, New York
  - Mountainview Medical Center, Berlin Corners, Vermont
  - Vermont Cancer Center, Burlington, Vermont
  - Vermont Center for Cancer Medicine, Colchester, Vermont

REFERENCES:
- [Derived] Moukharskaya J, Abrams DM, Ashikaga T, Khan F, Schwartz J, Wilson K, Verschraegen C, Openshaw T, Valentine J, Eneman J, Unger P, Ades S. Randomized phase II study of loratadine for the prevention of bone pain caused by pegfilgrastim. Support Care Cancer. 2016 Jul;24(7):3085-93. doi: 10.1007/s00520-016-3119-0. Epub 2016 Feb 19. PMID 26894485